CLINICAL TRIAL: NCT03878316
Title: Randomized, Double Blind, Placebo-Controlled Trial of the Efficacy of Intranasal Oxytocin for the Treatment of Alcohol Use Disorder
Brief Title: Intranasal Oxytocin for the Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCIG 007
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Alcohol Misuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Oxytocin (Active Comparator): Oxytocin, 35 IU per dose, intranasally twice-daily. One dose is defined as intranasal spray of 100 μL per each nostril x 5 sprays in alternating nostrils with a 30 second wait between sprays for a total dose volume of 500 μL. The total daily dose of oxytocin will be 70 IU/mL.
  Interventions: Drug: Instranasal Oxytocin
- Instrasal Placebo (Placebo Comparator): Identically matched placebo administered intranasally twice-daily. One dose is defined as intranasal spray of 100 μL per each nostril x 5 sprays in alternating nostrils with a 30 second wait between sprays for a total dose volume of 500 μL.
  Interventions: Drug: Instranasal Oxytocin

INTERVENTIONS:
Drug: Instranasal Oxytocin — Intranasal Oxytocin - concentrated formulation - 35 IU per dose

SUMMARY:
Primary: The primary objective of the study is to compare the efficacy of intranasal oxytocin in reducing the weekly percentage of heavy drinking days over the 10 weeks of maintenance treatment among subjects with moderate to severe Alcohol Use Disorder (AUD). A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.

Secondary: Secondary objectives include assessment of other measures of the effects of oxytocin compared with placebo on reduction of alcohol use as well as effects on psychological assessments, alcohol craving, alcohol-related consequences, cigarette smoking and other nicotine use, retention in the study, safety, and application site (nares) tolerability throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 21 years of age.
2. Have a current (past 12 months) DSM-5 diagnosis of AUD (4 or more symptoms) assessed using the MINI neuropsychiatric interview version 7.0.2 (at least moderate severity, ICD-10-CM Code F10.20 alcohol dependence, uncomplicated).
3. Have a BAC by breathalyzer equal to 0.000 when s/he signed the informed consent document (either just prior to or immediately after signing consent).
4. Be seeking treatment for problems with alcohol reduction in drinking.
5. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
6. Agree (if the subject is female and of child bearing potential) to use at least one of the following methods of birth control, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal:

   1. oral contraceptives,
   2. contraceptive sponge,
   3. patch,
   4. double barrier (diaphragm/spermicidal or condom/spermicidal),
   5. intrauterine contraceptive system,
   6. etonogestrel implant,
   7. medroxyprogesterone acetate contraceptive injection,
   8. complete abstinence from sexual intercourse, and/or
   9. hormonal vaginal contraceptive ring.
7. Be able to take intranasal investigational products and be willing to adhere to the investigational product regimen.
8. Complete all assessments required at screening and baseline.
9. Have a place to live in the 2 weeks prior to randomization and not be at risk that s/he will lose his/her housing by Study Week 14.
10. Not anticipate any significant problems with transportation arrangements or available time to travel to the study site by Study Week 14.
11. Not have any plans to move within Study Week 14 to a location which would make continued participation in the study impractical.
12. Not have any unresolved legal problems that could jeopardize continuation or completion of the study.
13. Provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the subject in case of a missed clinic appointment.
14. Be someone who in the opinion of the investigator would be expected to complete the study protocol.
15. Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may substantially interfere with study participation.
16. If taking a medication for depression or anxiety, must have been taking a stable dose in the 2-months prior to randomization and plan to continue during the study. This includes drugs such as the following:

    * SSRIs
    * Dual uptake inhibitors
    * SNRIs
    * Tricyclic antidepressants
    * MAOIs
    * Bupropion
17. Not currently taking oxytocin and agree not to take non-study oxytocin for the duration of the study.

Exclusion Criteria:

Contact study site for exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Litten, PHD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (4):
- United States (4):
  - University of California, Los Angeles, California
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Started | 50 | 50
Completed | 43 | 42
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes randomized participants who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin | Instrasal Placebo | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (10.8) | 51.1 (10.1) | 50.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 28 | 30 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 42 | 46 | 88
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 39 | 42 | 81
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
Percentage of heavy drinking days [Mean (Standard Deviation); unit: percentage of days] | 74.7 (23.0) | 79.8 (21.5) | 77.2 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Weekly Percentage of Heavy Drinking Days
Description: The primary efficacy endpoint is the weekly percentage of heavy drinking days during the 10-week maintenance treatment period. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men. Drinking data will be collected by the Timeline Followback (TLFB) method.
Time Frame: Weeks 3-12
Population: Full Analysis Set - randomized and received study medication
Measure: Least Squares Mean (Standard Error); unit: percentage of days per week
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
percentage of days per week | 51.5 (3.9) | 52.9 (3.9)

2. Secondary Outcome: Percentage of Subjects With no Heavy Drinking Days
Description: Percentage of subjects with no heavy drinking days during the 10-week Maintenance period
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Number; unit: percentage of participants
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
percentage of participants | 2.1 | 6.3

3. Secondary Outcome: Percentage of Subjects Abstinent From Alcohol
Description: Percentage of subjects abstinent from alcohol during the 10-week Maintenance period
Time Frame: Weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Number; unit: percentage of participants
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
percentage of participants | 0 | 2.1

4. Secondary Outcome: Percentage of Subjects With at Least a 1-level World Health Organization (WHO) Drinking Risk Category Decrease
Description: Percentage of subjects with at least a 1-level World Health Organization (WHO) drinking risk category decrease from the baseline level to (the period including the 28 days before screening) to the level during the treatment phase (Study Weeks 3-12).
  The WHO levels of average alcohol consumption per day vary by Sex of participants and are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g where 14g = 1 SDU (WHO-2000). In computing the WHO alcohol consumption level, average drinks per day were used, computed as the sum of all drinks in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects were included in a separate "Abstinent" category.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received study medication
Measure: Number; unit: percentage of participants
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
percentage of participants | 59.6 | 53.2

5. Secondary Outcome: Percentage of Subjects With at Least a 2-level World Health Organization (WHO) Drinking Risk Category Decrease
Description: Percentage of subjects with at least a 2-level World Health Organization (WHO) drinking risk category decrease from the baseline level to (the period including the 28 days before screening) to the level during the treatment phase (Study Weeks 3-12).
  The WHO levels of average alcohol consumption per day vary by Sex of participants and are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g where 14g = 1 SDU (WHO-2000). In computing the WHO alcohol consumption level, average drinks per day were used, computed as the sum of all drinks in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects were included in a separate "Abstinent" category.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received study medication
Measure: Number; unit: percentage of participants
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
percentage of participants | 23.4 | 23.4

6. Secondary Outcome: Percentage of Days Abstinent Per Week
Description: Timeline Follow Back daily drinking data used to calculate the % of days abstinent per week during the 10-week Maintenance period.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received study medication
Measure: Least Squares Mean (Standard Error); unit: percentage of days per week
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
percentage of days per week | 23.2 (2.5) | 22.6 (2.5)

7. Secondary Outcome: Weekly Mean Number of Drinks Per Week
Description: Weekly mean number of drinks per week during the 10-week Maintenance period.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: standard drinking units (SDUs) per week
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
standard drinking units (SDUs) per week | 33.1 (2.2) | 34.7 (2.3)

8. Secondary Outcome: Weekly Mean Drinks Per Drinking Day
Description: Weekly mean drinks per drinking day during the 10-week Maintenance period.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: standard drinking units (SDUs) per week
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
standard drinking units (SDUs) per week | 6.2 (0.3) | 6.3 (0.3)

9. Secondary Outcome: Number of Alcohol Use Disorder Symptoms (MINI)
Description: The MINI (paper version 7.0.2) is a short structured diagnostic interview, developed jointly by psychiatrists and clinicians in the United States and Europe, for DSM-5 and ICD-10 psychiatric disorders (Sheehan-1998). This scale is a count of the number of alcohol use disorder symptoms. Minimum = 0 and maximum=11. Higher scores indicate worse outcome.
Time Frame: week 13
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: Number of alcohol use disorder symptoms
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
Number of alcohol use disorder symptoms | 3.9 (0.3) | 4.2 (0.3)

10. Secondary Outcome: Cigarettes Smoked Per Week Among Smokers
Description: Cigarettes smoked per week among smokers during the 10-week Maintenance period.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Mean (Standard Deviation); unit: number of cigarettes smoked per week
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 4 | 7
number of cigarettes smoked per week | 40.6 (32.1) | 45.9 (52.8)

11. Secondary Outcome: Abstinence From Cigarette Smoking Among Smokers
Description: Abstinence from cigarette smoking among smokers during the 10-week Maintenance period.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Number; unit: percentage of participants
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 4 | 7
percentage of participants | 0 | 0

12. Secondary Outcome: Other Nicotine Product Use - Days Per Week Among Other Nicotine Product Users
Description: Other nicotine product use - days per week among other nicotine product users during the Maintenance period
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 4 | 8
days per week | 4.9 (1.9) | 5.4 (2.3)

13. Secondary Outcome: Experiences in Close Relationships-Relationship Structures Questionnaire (ECR-RS) Scores (Attachment-related Anxiety Subscale)
Description: Experiences in Close Relationships-Relationship Structures Questionnaire (ECR-RS) scores (attachment-related anxiety subscale) during the 10-week Maintenance period. Minimum = 0 and maximum = 126. Higher scores are worse outcome.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
score on a scale | 2.4 (0.1) | 2.4 (0.1)

14. Secondary Outcome: PROMIS Sleep Disturbances Score
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) Sleep Disturbances score (Short Form 8b) during the 10-week Maintenance period. Scores are T-scores with a mean of 50 and standard deviation of 10. Minimum = 0 and maximum = 100. Higher scores are worse outcome (i.e., more sleep disturbance).
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received study medication
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
T-score | 51.0 (0.7) | 51.3 (0.7)

15. Secondary Outcome: PROMIS Alcohol-related Negative Consequences Score
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) alcohol-related negative consequences score (Long Form) during the 10-week Maintenance period. Scores are T-scores with a mean of 50 and standard deviation of 10. Minimum = 0 and maximum = 100. Higher scores are worse outcome (i.e., more alcohol-related negative consequences).
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
T-score | 48.5 (0.6) | 47.7 (0.6)

16. Secondary Outcome: PROMIS Pain Interference Score
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) Pain Interference score (Short Form 8a) during the 10-week Maintenance period. Scores are T-scores with a mean of 50 and standard deviation of 10. Minimum = 0 and maximum = 100. Higher scores are worse outcome (i.e., more pain interference).
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
T-score | 52.2 (1.0) | 52.5 (1.0)

17. Secondary Outcome: Profile of Moods States (POMS) - Total Mood Disturbance
Description: Profile of Moods States (POMS) - Total Mood Disturbance during the 10-week Maintenance period. Minimum = -32 and maximum = 200. Higher scores are worse outcome.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
score on a scale | 8.9 (2.4) | 7.6 (2.4)

18. Secondary Outcome: Urge to Drink Alcohol Craving Score
Description: Urge to Drink alcohol craving score during the 10-week Maintenance period. Minimum = 0 and maximum = 35. Higher scores are worse outcome.
Time Frame: weeks 3-12
Population: Full Analysis Set - randomized and received medication
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
Number analyzed (Participants) | 49 | 48
score on a scale | 13.6 (0.7) | 13.2 (0.7)

ADVERSE EVENTS:
Time Frame: AEs were assessed at study visits starting after the first administration of investigational product (Day 1) until the final follow-up visit (Week 15). However, SAEs were collected from the time of informed consent (Day -14) until Week 15.
Description: General symptoms were collected via an open ended question: "How have you been feeling since your last clinic visit or phone contact?"?"
Arm/Group | Intranasal Oxytocin | Instrasal Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 44/49 | 45/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Oxytocin (N=49) | Instrasal Placebo (N=48)
Bradycardia (Cardiac disorders) | 4 (5) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Mucosal haemorrhage (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Pain and discomfort NEC (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Secretion discharge (General disorders) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (9) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (8) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 4 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine decreased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 2 (3)
Weight increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Food craving (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (7) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 6 (8) | 8 (10)
Hyposmia (Nervous system disorders) | 27 (45) | 25 (44)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (4) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (6)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 13 (35) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03878316/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03878316/SAP_001.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03878316/ICF_002.pdf